CLINICAL TRIAL: NCT05824884
Title: Self-efficacy Enhancement in a Virtual Reality Training for Fear of Heights: Promoting Mastery Experiences
Brief Title: Self-efficacy Enhancement in a Virtual Reality Training for Fear of Heights
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Armin Zlomuzica, Principal Investigator, Ruhr University of Bochum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AZ 794
Record Dates: First submitted 2023-04-08; First posted 2023-04-24 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Fear of Heights; Specific Phobia, Situational
Keywords: Specific phobia; fear of heights; Self-efficacy; virtual reality; exposure
MeSH Terms: conditions — Acrophobia; Phobia, Specific | interventions — Feedback, Sensory

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental 1 (Experimental): positive visual feedback during VR-height-exposure combined with SE-enhancement after exposure.
  Interventions: Behavioral: Visual Feedback; Behavioral: Self-efficacy enhancement:
- Active Comparator 1 (Active Comparator): positive visual feedback during VR-height-exposure, and a placebo intervention after exposure.
  Interventions: Behavioral: Visual Feedback; Behavioral: placebo intervention
- Active Comparator 2 (Active Comparator): no visual feedback during exposure but SE-enhancement after exposure.
  Interventions: Behavioral: Self-efficacy enhancement:; Behavioral: No visual feedback
- Placebo Comparator (Placebo Comparator): no visual feedback during exposure and placebo intervention after exposure.
  Interventions: Behavioral: placebo intervention; Behavioral: No visual feedback

INTERVENTIONS:
Behavioral: Visual Feedback — Visual progress feedback and words of positive affirmation will be presented triggered by checkpoints set in the VR-height-exposure.
  Arms: Active Comparator 1; Experimental 1
Behavioral: Self-efficacy enhancement: — specific instructions regarding the retrieval of mastery experiences during exposure will be given (modified version of the procedure used in Raeder et al. 2019).
  Arms: Active Comparator 2; Experimental 1
Behavioral: placebo intervention — specific instructions regarding the retrieval of the exposure session will be given without an emphasis on personal mastery experience (modified version of the procedure used in Raeder et al. 2019).
  Arms: Active Comparator 1; Placebo Comparator
Behavioral: No visual feedback — Participants can not trigger any checkpoints during VR and therefore not receive any progress feedback or positive affirmation.
  Arms: Active Comparator 2; Placebo Comparator

SUMMARY:
Self-efficacy (SE) enhancement after virtual reality exposure (VRET) for heights can promote treatment-induced effects (Raeder et al. 2019). Raeder et al (2019) employed an intervention to enhance SE by introducing specific questions about autobiographical events of success and mastery experiences in the course of VRET. Building on these previous findings, the present study aims to examine whether SE-enhancement DURING and/or AFTER a brief VR-based exposure for fear of heights (in the following referred to as VR-height-exposure) is suitable to promote exposure-induced reductions in height-related fear and avoidance. To this end, repeated visual feedback DURING a brief VR-height-exposure will be used to selectively promote SE and mastery experiences. In a similar vein, SE-enhancement AFTER VR-height-exposure will be administered. The effects of these interventions will be assessed on different treatment outcome levels. It will be further examined whether the combined SE enhancement (DURING and AFTER exposure) is more effective that 1.) SE enhancement performed DURING VR-height-exposure only or 2.) SE enhancement performed AFTER VR-height-exposure only.

The investigators hypothesize that SE enhancement (either administered DURING or AFTER VR-height-exposure) will be more effective (as indicated by more pronounced reductions in height-related fear and avoidance) than VR-height-exposure alone. It is further expected that the combined SE enhancement DURING and AFTER VR-height-exposure will be more effective compared to SE enhancement DURING VR-height-exposure alone and/or SE enhancement DURING VR-height-exposure alone.

DETAILED DESCRIPTION:
The aim of this study is to evaluate whether visual feedback DURING VR-height-exposure and SE-enhancement strategies that are designed to promote mastery experience AFTER exposure are suitable to benefit exposure-induced reductions in height-related fear and avoidance.

Participants will be randomly assigned to one of the following conditions: a) visual feedback DURING VR-height-exposure and SE-enhancement targeting mastery experience AFTER VR-height-exposure b) no visual feedback DURING VR-height-exposure but SE-enhancement targeting mastery experience AFTER VR-height-exposure, c) visual feedback DURING VR-height-exposure but a control intervention AFTER VR-height-exposure d) no visual feedback and control intervention after VR-height- exposure. The SE-enhancement as well as the control intervention involve memory reactivation either with or without emphasis on a mastery experience attained during the VR-height-exposure. The visual feedback is presented in form of a progress-update combined with positive affirmation.

The VR-height-exposure concludes different exercises in a virtual environment that simulate situations, that can be challenging to height-fearful individuals in real life, such as glass-elevators, a glass-bridge, a tall ladder and lattice stairs. During VR-height-exposure, self-reported fear is measured in Subjective Units of Distress (SUDS). The VR-environment is presented via head-mounted displays and the participants can use touch-controllers to navigate through the exercises guided by the experimenter.

As outcome measures, subjective fear and height-related avoidance will be assessed at three time points: pre-exposure, post-exposure and at 3 months-follow-up.

Subjective fear is measured using the Acrophobia Questionnaire (AQ; Cohen, 1977). To measure height-related avoidance behavior, a Behavioural Approach Test (BAT) will be performed in a nearby church tower, that includes 13 steps of varying difficulty and requires active behavioral approach towards height-situations.

Furthermore, danger expectancies and fear expectancies (DES, AES) will be measured at pre- and post-exposure as well as at 3-months-follow-up. During all BATs and the VR-height-exposure, heart-rate variability (HRV) will be assessed as a psychophysiological indicator for fear response.

Moreover, participants are asked to rate their general self-efficacy via Questionnaire (GSE) and their perceived self-efficacy via Visual Analogue Scales (VAS) at pre- and post-exposure as well as 3-months follow-up. Furthermore, the VAS measures mood, excitement, and distraction.

Additionally, several control variables are assessed pre-exposure, including Beck's Depression Inventory II (BDI-II), The State-and-Trait-Anxiety Inventory (STAI-T; STAI-S), the Self-Efficacy Scale (SES) and the CSSES.

Implicit Approach-Avoidance biases towards height-related stimuli will also be assessed pre- and post VR-height-training utilizing the Approach-Avoidance-Task (AAT). The participants are instructed to push away (simulating avoidance) vs. pull towards (simulating approach) neutral vs. height-related pictures according to the way they are tilted (tilted-right vs. tilted left) using the computer mouse. Reaction time delays in the pull towards height-related pictures condition can be an indicator for implicit avoidance tendencies.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 65 years
* fear of heights
* normal or corrected vision

Exclusion Criteria:

* acute psychotherapy or psychotherapy in the past 2 years
* acute psychiatric drug intake
* acute schizophrenic or psychotic symptoms
* acute major depressive episode with severe symptoms
* acute substance use disorder
* neurological disorder or mental disability
* cardiac arrhythmias or pacemaker

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-06-22 (Actual); Primary Completion 2026-03-03 (Estimated); Study Completion 2026-03-03 (Estimated)

PRIMARY OUTCOMES:
Change in the Behavioural Approach Test (BAT) | from baseline to 24 hours after exposure and 3-months-follow-up
Change in Acrophobia Questionnaire (AQ) | from baseline to 24 hours after exposure and 3-months-follow-up
Change in subjective fear during the BAT | from baseline to 24 hours after exposure and 3-months-follow-up
  Subjective fear during the BATs will be measured using the Subjective Units of Distress Scale (SUDS)
Changes in Heart Rate Variability (HRV) during the BAT | at baseline, 24 hours after exposure and at 3-months-follow-up

SECONDARY OUTCOMES:
Change in Danger Expectancy Scale (DES) | from baseline to 24 hours after exposure and 3-months-follow-up
Change in Anxiety Expectancy Scale (AES) | from baseline to 24 hours after exposure and 3-months-follow-up
Differences in GSE between the respective groups | at pre-exposure, immediately after exposure and 3-months-follow-up
  ANOVA with mean GSE-scores
Differences in AQ between the respective groups | at baseline, 24 hours after exposure and 3-months-follow-up
  ANOVA with mean AQ-scores

OTHER OUTCOMES:
Change in perceived SE from pre to post VR-height-exposure | from baseline to 24 hours after exposure and 3-months-follow-up
  Changes in perceived SE will be measures with visual analogue scales (VAS)
Becks Depression Inventory II (BDI) | assessed at baseline
State-Trait Anxiety Inventory (STAI-T/STAI-S) | assessed at baseline
Self-Efficacy Scale (SES) | assessed at baseline
Chronic Stress Self-Efficacy Scale (CSSES) | assessed at baseline
Avoidance Bias in height-fearful individuals | assessed at baseline
  An Avoidance Bias will be assessed utilizing the AAT
Changes in Avoidance Bias | from baseline to 24 hours after exposure

CONTACTS AND LOCATIONS:
Locations (1):
- Mental Health Research and Treatment Center, Bochum, Germany